CLINICAL TRIAL: NCT04361955
Title: Modulatory Effects of Deep Brain Stimulation on Cerebral Cortical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Farmer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-028
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: DBS; Parkinson Disease; Essential Tremor; Healthy
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Intervention Model Description: Study N = 180 participants 60 participants with diagnosis of essential tremor having DBS implanted 70 participants with diagnosis of Parkinson Disease having DBS implanted 50 healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- PD with DBS on (Other): intervention is EEG while at rest and performing tasks, on anti PD medications and off anti PD medications
  Interventions: Other: EEG
- PD with DBS off (Other): intervention is EMG while at rest and performing tasks, on anti PD medications and off anti PD medications
  Interventions: Other: EMG
- ET with DBS on (Other): intervention is EEG while performing tasks and at rest
  Interventions: Other: EEG
- ET with DBS off (Other): intervention is EEG while performing tasks and at rest
  Interventions: Other: EMG

INTERVENTIONS:
Other: EMG — recordings of muscle electrical activity during nerve stimulation using EMG
  Arms: ET with DBS off; PD with DBS off
Other: EEG — recordings of brain activity using EEG
  Arms: ET with DBS on; PD with DBS on

SUMMARY:
The purpose of this study is to learn about how deep brain stimulation (DBS) affects brain activity in those with Parkinson's disease (PD) and essential tremor (ET). The effect of therapeutic and non-therapeutic stimulation settings will be assessed. Additionally, DBS effects in the presence and absence of anti-PD medication will be studied. Also of interest are differences in stimulation effects while at rest versus while performing a task.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is a standard-of-care, FDA approved therapy for Parkinson's disease (PD) and tremor and well over 1,000 patients have been implanted at the Cleveland Clinic in the past 20 years. The therapy involves stereotactic implantation of one or more leads into specific sensorimotor brain regions, with each lead consisting of an array of four to eight contacts. The proximal end of the lead is tunneled to an implantable pulse generator (IPG) placed under the skin of the chest. Post-operatively, a health care professional carefully programs the IPG: adjusting the delivery location (i.e., contact selection) and titrating the frequency, amplitude, and width of the stimulus pulses to maximize therapeutic benefit while minimizing any side effects. It is hypothesized that the chronic, electrical stimulation of the target region has both local and circuit-wide effects, the net effect of which is to disrupt the pathophysiological neural activity present across both cortical and subcortical brain regions that is thought to underlie disease manifestation.

Study-related activities will begin in the morning, with participants reporting to the Center for Neurological Restoration outpatient clinic desk in the S-building. Those participants with a diagnosis of Parkinson's disease will be asked to arrive in the "practically defined OFF" state (i.e., will come for testing having taken PD medications as usual up to midnight of the preceding day, and none on the morning of testing). To help to minimize off-medication risks, patients with PD will be offered the option to stay overnight at an on-campus hotel at no cost. Patients will be provided with lunch and additional rest breaks, as needed, throughout the day.

A technician will apply either Ag/AgCl clinical scalp electrodes or an elastic cap pre-populated with electrodes after which electroencephalographic (EEG) activity will be monitored and recorded throughout the remainder of the study. Participants will undergo an initial stimulation threshold evaluation to establish DBS-related sensorimotor side effect thresholds.

Throughout testing, participants will be seated comfortably in a quiet room. Continuous EEG and EMG recordings will be made as the parameters of the patients IPG are systematically modified (i.e., changes in pulse frequency, amplitude, width and active contacts) with the patient at rest and, for specific settings, again while the patient performs a simple, continuous motor task using the upper extremity (e.g., computer-generated sine tracking). Visual and auditory evoked potentials will be elicited using stimuli delivered via goggles (or other light source) and headphones, respectively. Somatosensory evoked potentials will be elicited through electrical stimulation of the median or posterior tibialis nerve using standard clinical techniques at approximately 125% of motor threshold. Event related potentials tasks will include simple and choice reaction time, NoGo, as well as auditory oddball tasks repeated in one or more DBS conditions. Note that the precise order of test administration may be randomized in order to minimize order effects. Also note that patients diagnosed with PD will be instructed to take their usual dose of anti-PD medication approximately mid-way through the test session, after which a subset of the evoked potential testing will be repeated.

In this study, the investigators will use multiple non-invasive physiological metrics, including scalp electroencephalography and surface electromyography, to characterize the spatiotemporal pattern of cortical and corticomuscular modulation associated with therapeutic, non-therapeutic, and side-effect-inducing parameters of DBS to address the specific aims.

ELIGIBILITY:
Inclusion Criteria:

* between 40 and 80 years old
* ability to consent
* diagnosis of idiopathic Parkinson Disease or ET for a duration of at least 4 years
* implanted with DBS (STN, GPi or VIM) for at least 3 months

Exclusion Criteria:

* secondary Parkinsonism, stroke, or progressive central nervous system disease other than Parkinson's disease or essential tremor
* cognitive impairment meeting criteria for dementia on formal neuropsychological evaluation
* lack of fluency in English which would invalidate cognitive testing
* current alcohol or substance abuse
* hearing or visual impairment precluding sensory or cognitive testing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
characterize and record brain activity | collected during the 8 hour office visit
  1) Characterize the spatial and temporal characteristics of cortical activity evoked in response to deep brain stimulation of the targeted subcortical nucleus. 2) Determine the effect of dopamine replacement therapy (DRT) on the spatial and temporal characteristics of the evoked cortical potentials (PD Patients only). 3) Determine the effect of patient state (rest vs. active) spatial and temporal characteristics of the evoked cortical potentials.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Baker, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States